CLINICAL TRIAL: NCT06368973
Title: Mechanical Ventilation-Associated Complications and Co-Morbidities in Children Admitted in Pediatric Intensive Care Unit: A Retrospective Study
Brief Title: Mechanical Ventilation-Associated Complications and Co-Morbidities in Children Admitted in Pediatric Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amany Mohammed El-Rebigi, MD, Lecturer of Pediatric and Neonatology, Benha University
Other Study IDs: RC16-4-2023
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Mechanical Ventilation Complication
Keywords: Mechanical Ventilation, Complications,Co-morbidities.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study was to identify the prevalence of mechanical ventilation-associated complications and co-morbidities in pediatric patients admitted to the PICU of Benha University Hospital, uncover how often these problems occur, their types, factors linked to them and to compare the epidemiology of MV-associated complications.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is used frequently for critically ill children in pediatric intensive care unit (PICU). While respiratory disease is a major indication for invasive mechanical ventilation (IMV), there are also numerous non-respiratory indications for mechanical ventilation, including neurological and neuromuscular pathology, congenital heart disease, hemodynamic shock, and postoperative care and pain management and septic shock.

Although lung-protective ventilation strategies are extensively implemented in the pediatric population, frequent adverse events (AEs) of mechanical ventilation are detected, such as accidental extubation, atelectasis, trauma by aspiration, ventilator-associated pneumonia (VAP), perioral tissue damage, secretion-mediated obstruction of the endotracheal tube (ETT), mucus plugging, air leak syndromes, neuromyopathy, post-extubation stridor, and PICU delirium. Some of these events require the direct intervention of the physician, nurse, or physiotherapist in order to be identified; thus, they are associated with the quality of care.The incidence of these complications among pediatric patients in the PICU is noteworthy, with rates ranging from 27 to 97 adverse events per thousand patients per day. This is mainly associated with hazardous invasive procedures that can lead to unfortunate poor outcome.Few studies focus on the complications of using ventilators in infants and adolescents, especially regarding VAP cases.

The goal of this study was to identify the prevalence of mechanical ventilation-associated complications and co-morbidities in pediatric patients admitted to the PICU of Benha University Hospital, uncover how often these problems occur, their types, factors linked to them and to compare the epidemiology of MV-associated complications.

ELIGIBILITY:
Inclusion Criteria:

* all pediatric patients aged 29 days to 16 years who were admitted to the pediatric intensive care unit and underwent invasive mechanical ventilation for at least 24 hours between January 2021 and December 2023.

Exclusion Criteria:

* newborns (<29 days old),
* pediatric patients received invasive mechanical ventilation less than 24 hours
* children with chronic respiratory failure or unable to be discharged due to socioeconomic constraints and requiring long-term mechanical ventilation therapy and pediatric patients with incomplete data or transferred to another hospital.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all pediatric patients aged 29 days to 16 years who were admitted to the PICU and underwent IMV for at least 24 hours between January 2021 and December 2023. Our analysis included data gathered from the follow-up medical records maintained by the PICU team and other healthcare providers.
Sampling Method: Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse events associated with mechanical ventilation | 4 weeks after following usage of invasive mechanical ventilation
  to assess incidence of complications associated with invasive ventilation in critically ill children

CONTACTS AND LOCATIONS:
Overall Officials: Amany M. El-Rebigi, MD, Principal Investigator — Pediatric and Neonatology Department, Benha Faculty of Medicine, Benha University, Benha, Egypt
Locations (1):
- Benha University Hospital, Cairo, Egypt